CLINICAL TRIAL: NCT05396781
Title: Acceptability and Performance of a Mobile Optical Biopsy Technology for Gastrointestinal Cancer Screening: A Clinical Study in Brazil
Brief Title: Acceptability and Performance of a Mobile Optical Biopsy Technology for Gastrointestinal Cancer Screening
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anandasabapathy, Sharmila, M.D. (Individual)
Collaborators: William Marsh Rice University (Other); Baylor College of Medicine (Other); University of Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-44015
Record Dates: First submitted 2022-02-11; First posted 2022-05-31 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Suspected or Known Squamous Cell Neoplasia; Prior History of Squamous Cell Dysplasia and /or Neoplasia
Keywords: Squamous cell neoplasia; Proflavine; Lugol's chromoendoscopy
MeSH Terms: conditions — Neoplasms | interventions — Proflavine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Augmented Reality High Resolution Microendoscope (HRME) imaging (Experimental): All study subjects will receive White Light Imaging and Lugol's Chromoendoscopy (LCE) which is the current standard of care procedure. The investigators will record any LCE abnormal areas and record the clinician's plan of action. Following LCE, all subjects will receive Mobile, Augmented Reality High Resolution Microendoscope (marHRME) imaging with the study contrast agent (Proflavine) of any LCE-identified abnormal areas as well as LCE normal areas. The investigators will record the subjective clinician read and confidence level in the investigators' diagnosis, and plan of action. Then the investigators will image the same abnormal and normal areas with the marHRME and record the software read, clinician confidence level, and plan of action. Finally, the imaged areas will be biopsied or resected and evaluated by a pathologist. All subjects will receive both standard of care and marHRME imaging.
  Interventions: Drug: Proflavine; Device: Mobile, Augmented High Resolution Microendoscope

INTERVENTIONS:
Drug: Proflavine — 5-10 ml of proflavine hemisulfate (0.01%) will be sprayed on the esophageal mucosa.
  Other Names: proflavine hemisulfate
Device: Mobile, Augmented High Resolution Microendoscope — The marHRME will then be inserted through the endoscope and gently placed against the mucosa. Imaging of abnormal tissues will be performed.
  Other Names: marHRME

SUMMARY:
The investigators have a current trial in China and the US which provides significant support for the safety, cost-effectiveness, accuracy and efficiency of a high resolution microendoscope (HRME)-guided approach in the hands of experienced clinicians. To improve functionality, portability and broader use of this device by non-experts, the investigators recently developed a prototype marHRME platform with an automated, augmented reality (AR)-interpretation that provides an overlaid endoscopic + micro-endoscopic view, facilitating diagnosis and biopsy targeting.

DETAILED DESCRIPTION:
The investigators' hypothesis is that this mobile device with automated, AR optical biopsy diagnoses can efficiently and accurately facilitate endoscopic cancer detection in low to middle income countries (LMICs) with less experienced providers and is acceptable to providers and patients.

Objective 1: The investigators' first objective is to evaluate the marHRME technology in terms of performance, efficiency, and impact. In a single-arm, feasibility study (n=50) of high-risk subjects undergoing Lugol's chromoendoscopy (LCE) followed by marHRME for esophageal squamous cell neoplasia (ESCN) screening, the investigators will evaluate the diagnostic performance and efficiency of this automated optical biopsy device.

The investigators' main hypothesis is that the marHRME will:

1. increase the accuracy of Lugol's endoscopy (LCE), other exploratory hypotheses are
2. increase the accuracy of marHRME among novices and be non-inferior to experts,
3. increase user confidence among experts and novices and, subsequently,
4. increase the efficiency and impact of LCE by reducing biopsies and second procedures.

For performance for marHRME vs. Standard of Care, the investigators will compare the accuracy of the marHRME + LCE vs. LCE alone to the gold-standard histopathology (expert GI pathologist). For performance of the Machine vs. Man, the investigators will compare accuracy of the marHRME software read to novice and expert clinicians' subjective read to gold-standard histopathology. For clinician confidence and clinical impact, the investigators will determine the clinician's confidence level in the software diagnosis and the potential clinical impact of this diagnosis among novice and expert endoscopists using marHRME.

Objective 2: The investigators' secondary objective is to evaluate the acceptability of the technology among patients and providers. All patients participating in the study will be invited to participate in a brief (20 min) interviewer-administered survey prior to undergoing endoscopy to assess attitudes and barriers to marHRME, and a follow-up interview (7 days post-procedure) to determine experiences and acceptability. Informed consent and the initial interview will be conducted in a private clinic room by trained study staff from the Brazilian team using a brief Portuguese-language survey. The follow-up interview will occur by phone, after a routine follow-up call by clinical staff.

The endoscopists and trainees participating in the feasibility study will be invited to participate in a series of questionnaires and in- depth interviews administered at different time points of the study to assess provider acceptance. Informed consent will be obtained prior to the first interview. Clinicians will answer a brief questionnaire to assess acceptance of marHRME prior to undergoing raining, after training, and after conducting 25 procedures. After 25 procedures, endoscopists and trainees will participate in a 30- minute semi-structured interview to assess marHRME experience. The interviews will be audio recorded, professionally transcribed, and translated (Portuguese to English) for coding and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients undergoing routine (standard of care) Lugol's chromoendoscopic screening for squamous cell neoplasia will be eligible for enrollment including patients with known history of head/neck squamous cell cancer.
* Patients must be >18 years old and able to give informed consent.
* For the provider surveys and interviews, all providers (clinicians, trainees) who are working on the project will be eligible to participate.

Exclusion Criteria:

* Allergy or prior reaction to the fluorescent contrast agent proflavine
* Patients who are unable to give informed consent
* Known advanced squamous cell carcinoma of the distal esophagus, or dyplastic/suspected malignant esophageal lesion greater than or equal to 2cm in size not amenable to endoscopic therapy
* Patient unable to undergo routine endoscopy with biopsy
* Women who are pregnant or breastfeeding
* Prothrombin time greater than 50% of control; Partial Thromboplastin Time greater than 50 sec, or International Normalized Ratio greater than 2.0
* inability to tolerate sedated upper endoscopy due to cardio-pulmonary instability or other significant medical issues
* Providers will be excluded if they decline participation or otherwise opt out of the proposed research project.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield | Day 1
  The number of neoplastic biopsies/total number of biopsies obtained in patients who received biopsies.
'Patient saved' | Day 1
  The number of patients who received no biopsies.
Procedure time | During Procedure
  Total procedure time added by the HRME imaging.

SECONDARY OUTCOMES:
Clinical impact | Day 1
  The number of cases that a change in clinician plan of action was noted from LCE interpretation only to LCE+HRME interpretation.

OTHER OUTCOMES:
Performance Characteristics | Day 1
  Comparison of accuracy of HRME to LCE for the prediction of squamous esophageal neoplasia using histopatholgy as the gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila Anandasabapathy, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- Baylor College of Medicine, Houston, Texas, United States
- University of Sao Paulo, São Paulo, São Paulo, Brazil

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT05396781/Prot_SAP_000.pdf